CLINICAL TRIAL: NCT05818501
Title: The Effectiveness and Feasibility of Dysphagia Cups in Elderly and Rehabilitation Setting: A Single Group Pre-post Test Study
Brief Title: Dysphagia Cups in Elderly and Rehabilitation Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Haven of Hope Hospital (Other); The Social Innovation and Entrepreneurship Development Fund, Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Derek Yee-Tak Cheung, Principal Investigator, Assistant Professor, The University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Care food_protocol_v2
Record Dates: First submitted 2023-04-04; First posted 2023-04-18 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Technology
Keywords: Gerontechnology; Risk; Water consumption; Autonomy

STUDY DESIGN:
Intervention Model Description: The trial is a single group pre-post test study at elderly residential settings and rehabilitation settings. During the 12-day or 13-day trial period, the participants will use conventional cups in the first 5 days of the trial, receive 2-3 days of training on using the one of the two models of dysphagia cups, and use the dysphagia cups for 5 days.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The dysphagia cups (Experimental): The participants will use the one of the two models of dysphagia cups for 5 days during trial period.
  Interventions: Device: The dysphagia cups

INTERVENTIONS:
Device: The dysphagia cups — After the training period of the one of dysphagia cups, participants will start using cup to consume water during a designated period of time every day.
  Participants consuming water with Cup A will drink from a static position with their chins towards their chests, the so-called Chin-Tuck maneuver. This position leads epiglottal naturally covering the trachea and causes liquid only ﬂowing to the esophagus and thus stomach. The restoring force of the membrane ensures a constant level of liquid at the upper edge of the cup and thus enables this preferred and safe drinking position.
  Cup B limits the maximum volume of water flowing out of the Cup B designated by the staff. Controlled liquid flow prevents overflowing the mouth and gulping, thus reduces the risk of choking and liquid aspiration. Participants can choose to drink the water from Cup B with a straw when necessary.

SUMMARY:
The study has 6 research questions regarding the use of dysphagia cups:

Primary study questions:

1. Can the use of the dysphagia cups increase water consumption and liquid consumption during the trial period?
2. Can the use of the dysphagia cups reduce the frequency and intensity of choking and coughing while drinking?
3. What are the potential risks to the service users while using the dysphagia cups?

   Secondary study question:
4. Can the use of the dysphagia cups enhance the autonomy of the service users in drinking?

   Auxiliary study questions:
5. Can the use of the dysphagia cups reduce the amount of thickener used for water consumption?
6. What are the perceived benefits and acceptability of using the dysphagia cups?

DETAILED DESCRIPTION:
Study design

The trial is a single group pre-post test study. During the 12-day or 13-day trial period, the participants will use conventional cups in the first 5 days of the trial, receive 2-3 days of training on using the one of the two models of dysphagia cups (Cup A and Cup B), and use the dysphagia cups for 5 days.

This protocol complies with the International Council for Harmonisation of Technical Requirements for Pharmaceuticals for Human Use - Guideline for Good Clinical Practice (ICH-GCP).

Procedures

1. Staff training

   For each of the drinking aid model, a few identical 60-min training sessions on sanitizing and preparing dysphagia cups (including resembling the cups, pouring water into the cups, positioning the cups so that service users can drink the water in the cups etc.) will be delivered to all related staff.
2. Participants' recruitment and consent

   The occupational therapist, speech therapist or the nurse of the service units will screen for and invite eligible service users to join the study.

   Service users scoring above the cutoff for dementia in Montreal Cognitive Assessment (MoCA) (see Appendix 1) and not receiving a medical diagnosis of dementia or other mentally incapacitating disease will be classified as competent in giving consent and will be invited to give consent.

   For elderly with dementia scoring below the cutoff in MoCA or receiving a diagnosis of mentally incapacitating disease, and persons in the rehabilitation setting, the criteria stated in the Alzheimer Europe Report (2011) will be followed to ensure that they are provided chances to give consent. In particular, four criteria will be evaluated, including 1) the person must have sufficient capacity to understand the information, 2) the person is able to retain, use and weight up such information for making a decision, 3) the person will understand the benefit, risk, and convenience, 4) the person must have the ability to communicate the decision. The University of Hong Kong (HKU) research staff and the care staff will first commit them in a causal chat to assess their ability to communicate and understand the dialogues.

   If service users are competent in giving consent, both service users and their next of kin will be approached for consent. In cases service users are not competent in giving consents, only their next of kin will be approached for consent. They will then be referred to join a 1-to-1 study introduction session. In this session, HKU research staff and service unit staff will introduce the study to the participant, and invite them to sign a consent form.

   For care staff, written informed consent will be obtained before doing qualitative interview.
3. Pre-test

   Before the use of the dysphagia cups, there will be 5-day pre-test. During the pre-test, participants will continue to use the conventional cup to drink water. To accurately record the volume of water consumption, service users from elderly residential settings will only consume water from a specific 2-litre jar. For service users from rehabilitation settings, they will consume water with conventional cups at the designated time (i.e., during breakfast, lunch and dinner). In this period, the care staff will complete a daily survey recording (1) the volume of water consumed by each participant at the designated time, (2) volume of liquid consumed by each participant every day during the pre-test period, (3) the frequency and intensity of choking and coughing while drinking, and (5) the autonomy of the participants in drinking measured by self-developed rating scale. (6) The amount of thickener used for water consumption will be retrieved from record.
4. Training period

   Following the pre-test, each participant will then receive cup training for 2 to 3 days. The responsible clinical staff will observe the selected training session(s) for potential risks and produce (4) the findings in an observation report. The report will be used to revise the operations protocol and for follow-up staff training.

   Participants consuming water with Cup A will drink from a static position with their chins towards their chests, the so-called Chin-Tuck maneuver. This position leads epiglottal naturally covering the trachea and causes liquid only ﬂowing to the esophagus and thus stomach. The restoring force of the membrane ensures a constant level of liquid at the upper edge of the cup and thus enables this preferred and safe drinking position.

   Cup B limits the maximum volume of water flowing out of the Cup B designated by the staff. Controlled liquid flow prevents overflowing the mouth and gulping, thus reduces the risk of choking and liquid aspiration. Participants can choose to drink the water from Cup B with a straw when necessary.
5. Formal testing period

After the training period, participants will start using the Cups to consume water during a designated period of time every day for 5 days. Fluids other than water, for example, soup, juice and milk, will be consumed using conventional cup, and their volume will also be recorded. Similar to the pre-test arrangement, service users from elderly residential settings will only consume water from the specific 2-litre jar whereas service users from rehabilitation settings will consume water with dysphagia cups at the designated time (i.e., during breakfast, lunch and dinner). Staff will prepare the dysphagia cups for the participants when needed. They will record the volume of water remaining in the jar throughout the formal testing period. After every meal, in case the participant does not drink enough liquid as perceived by the staff, the staff will try all means to encourage the participants to drink enough water, including using the conventional cups which will be the last resort. The volume of water consumed using conventional cups will be estimated by the staff based on the number of cups of water offered and estimated amount of water remaining.

In this period, the care staff will complete a daily survey recording (1) the volume of water consumed by each participant at the designated time, (2) volume of liquid consumed by each participant every day during the formal testing period, (3) the frequency and intensity of choking and coughing while drinking, and (5) the autonomy of the participants in drinking measured by self-developed rating scale. (6) The amount of thickener used for water consumption will be retrieved from record.

Qualitative interviews will be conducted with all participants who can communicate at the end of the formal testing period. 2-3 related staff of each site will be interviewed after all participants have completed or terminated the trial. Interview contents include the perceived benefits and feasibility in allowing the participants to the drinking aid(s) as compared to conventional cups.

Blinding

No blinding will be done for this single group study.

Sample size determination

The sample size is estimated by the expected number of eligible service users and the number of care staff responsible for helping them to drink water. It is estimated that a total of 12-30 service users and 8-30 care staff will be using the dysphagia cups.

Data analysis

1. Main analysis

   Independent sample t-test will be used to evaluate the difference in average daily water consumption, average daily liquid consumption, frequency and intensity of choking and coughing while drinking, the autonomy of the service users in drinking, and the amount of thickener used for water consumption.

   The observation reports regarding the potential risks will be summarized.
2. Qualitative interview

The content will be transcribed verbatim in Chinese for further analysis. Transcripts will be analysed using framework analysis to construct a coherent and logical structure from the classification of many opinions and perceptions of the new and conventional cups. The results will then be discussed and consolidated in the panel meetings with the co-authors.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for service users using Cup A:

* Is recommended to consume liquid at the International Dysphagia Diet Standardisation Initiative (IDDSI) level 1 or 2, by the speech therapist, occupational therapist or nurse of the study site,
* Able to perform chin-down posture when swallowing,
* Able to hold Cup A with single hand or both hands, and
* Able to understand Chinese

Inclusion criteria for service users using Cup B:

* Is recommended to consume liquid at the International Dysphagia Diet Standardisation Initiative (IDDSI) level 1 or 2, by the speech therapist, occupational therapist or nurse of the study site,
* Able to hold Cup B with single hand or both hands, or drinking water using straws, and
* Able to understand Chinese

Inclusion criteria for staff:

* Responsible for helping participants to drink water using conventional cups (i.e. occupational therapist, speech therapist, nurse and care staff), and
* Able to understand Chinese

Exclusion Criteria:

Exclusion criteria for service users using Cup A:

- Not able to learn to use Cup A during training session

Exclusion criteria for service users using Cup B:

- Not able to learn to use Cup B during training session

Exclusion criteria for staff:

- None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2023-07-13 (Actual); Primary Completion 2023-09-11 (Actual); Study Completion 2023-09-11 (Actual)

PRIMARY OUTCOMES:
Change of daily water consumption before and after using the dysphagia cup for 5 days | From the start of 5-day pre-test to the end of 5-day trial period
  Change of water consumption (including all sugar- and oil-free fluid) of each participant at the designated time in using the conventional cup for 5-day pre-test and the dysphagia cups for 5-day trial period will be recorded by the care staff every day. The volume value is expressed in the unit of milliliter.
Change of daily actual liquid consumption in using conventional cup and dysphagia cup | From the start of 5-day pre-test to the end of 5-day trial period
  Change of actual liquid consumption (including water consumption using both dysphagia cups and conventional cups and other liquid consumption, e.g. soup, milk and juice) of each participant will be recorded by the care staff every day from the pre-test period to the formal trial period. The volume value is expressed in unit of milliliter.
Change of frequency of choking and coughing every day before and after using the dysphagia cup | From the start of 5-day pre-test to the end of 5-day trial period
  Change of frequency of choking and coughing while drinking in using the conventional cup for 5-day pre-test and the dysphagia cup for 5-day trial period will be counted and recorded by the care staff every day.
Change of intensity of choking and coughing every day before and after using the dysphagia cup | From the start of 5-day pre-test to the end of 5-day trial period
  Change of intensity of choking and coughing while drinking in using the conventional cup for 5-day pre-test and the dysphagia cup for 5-day trial period will be observed and recorded by the care staff every day. Care staff will complete an item and the minimum and maximum values of scale is 0 and 2 respectively, with higher score indicating more choking and coughing while drinking.
Qualitative measures: Potential risks to service users while using the dysphagia cups | From the start to the end of 2- or 3-day training period
  During the training of each dysphagia cup, the responsible clinical staff will observe the selected training session(s) for potential risks and produce the findings in an observation report. The contents include resembling the cups, pouring water into the cups and positioning the cups.

SECONDARY OUTCOMES:
Change of autonomy of service users in drinking before and after using the dysphagia cup | From the start of 5-day pre-test to the end of 5-day trial period
  Change of autonomy of service users while drinking in using the conventional cup for 5-day pre-test and the dysphagia cup for 5-day trial period will be observed and recorded by the care staff every day. Care staff will complete an item on self-developed rating scale and the minimum and maximum values of the scale is 0 and 3 respectively, with the higher score indicating the higher level of autonomy.
Change of the amount of thickener used for water consumption before and after using the dysphagia cup | From the start of 5-day pre-test to the end of 5-day trial period
  Change of the amount of thickener used for water consumption with the conventional cup and the dysphagia cups will be retrieved form record by care staff.
Qualitative measures: The perceived benefits and acceptability of the dysphagia cups for participants | At the end of the 5-day trial period
  All participants who can communicate will be interviewed after all participants have completed or terminated the trial. Interview contents include:
  1. Do you like the appearance of the cup?
  2. Is it easy to use?
  3. Is it comfortable to consume water with the cup?
  4. Do you think the risk of choking and coughing can be reduced while drinking?
  5. Do you like/dislike the dysphagia cup?
  6. Do you want to continue to use the cup in the future?
Qualitative measures: The perceived benefits and acceptability of the dysphagia cups for caregivers | At the end of the 5-day trial period
  A total of 2-3 related staff of each site will be interviewed after all participants have completed or terminated the trial. Interview contents include:
  1. To compare with the conventional cup, do you think the appearance of the dysphagia cup can encourage service user to consume water?
  2. How is the size of dysphagia cup?
  3. Is it easy to assemble the cup?
  4. Were service users willing to use the cup?
  5. To compare with the conventional cup, did the frequency of choking or coughing can be reduced in using the dysphagia cup?
  6. Did you discover other benefits due to the use of the dysphagia cups?
  7. What were your concerns when you were asked the service users to use the cup?
  8. On the whole, are you satisfied with the cup?
  9. To what extent, do you want the service users to continue to use the cup?

CONTACTS AND LOCATIONS:
Overall Officials: Yee Tak Cheung, PhD, Principal Investigator — The University of Hong Kong
Locations (6):
- Hong Kong (6):
  - Haven of Hope Hang Hau Care and Attention Home for Severely Disabled, Hong Kong
  - Haven of Hope Ming Tak Day Activity Centre cum Hostel - Extended Care Programme, Hong Kong
  - Haven of Hope Sister Annie Skau Holistic Care Centre, Hong Kong
  - Haven of Hope Tsui Lam Day Care Centre for the Elderly, Hong Kong
  - Haven of Hope Woo Ping Care & Attention Home, Hong Kong
  - Haven of Hope Yee Ming Day Care Centre for the Elderly, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
Research data and documentation will be available upon request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be available for 10 years.